CLINICAL TRIAL: NCT02609165
Title: Nerve Growth Factor Eye Drops as a Novel Treatment for Vision Loss in Patients With Retinitis Pigmentosa: From Preclinical to Clinical Phase II Trial
Brief Title: Nerve Growth Factor Eye Drops Treatment in Patients With Retinitis Pigmentosa and Cystoid Macular Edema
Acronym: NEMO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Collaborators: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Principal Investigator, Paolo Rama, MD, Ospedale San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RF-2010-2318561
Record Dates: First submitted 2015-10-12; First posted 2015-11-20 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Retinitis Pigmentosa; Cystoid Macular Edema
MeSH Terms: conditions — Retinitis Pigmentosa; Macular Edema | interventions — cenegermin; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Active Comparator): rhNGF 180 µg/ml eye drops solution
  Interventions: Drug: rhNGF 180 µg/ml eye drops solution
- control group (Placebo Comparator): vehicle eye drops solution
  Interventions: Drug: vehicle eye drops

INTERVENTIONS:
Drug: rhNGF 180 µg/ml eye drops solution — eye drops
  Other Names: recombinant human Nerve Growth Factor
  Arms: study group
Drug: vehicle eye drops — placebo
  Other Names: vehicle eye drop solution
  Arms: control group

SUMMARY:
This study aims at investigating the therapeutic potential of recombinant human Nerve Growth Factor ( rhNGF ) eye drops treatment in patients with Retinitis Pigmentosa (RP) associated with cystoid macular edema (CME) in a phase II, randomized, double-masked, controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Typical and atypical forms of retinitis pigmentosa (RP)
2. Measurable ERG with a significant decrease in the amplitude .
3. Reduction of the visual field (assessed with Humphrey field analyzer- HFA 24-2) and values of mean deviation> -3 decibel (dB).
4. RP associated with CME documented by OCT (macular thickness greater than 250 uM) present for at least three months and not in treatment for at least one month;
5. Best corrected visual acuity (BCVA) between 20/100 (2/10 or 0.1 logMAR) and 20/25 (8/10 or 0.7 logMAR) and best corrected visual acuity for near not exceeding II character
6. Absence Other ocular confounding diseases
7. Participant must be medically able to undergo the testing and study procedures required in the flowsheet of exam procedures.

Exclusion Criteria:

1. Presence of diabetes-related macular edema, or macular edema associated with other causes such as choroideal neovascularization or after the eye surgery.
2. patients with diabetes mellitus.
3. Patients who have performed eye surgery in the previous three months.
4. Evidence of an active eye infection.
5. previous uveitis or evidence of intraocular inflammation.
6. History or evidence of glaucoma or elevated intraocular pressure (IOP) greater than or equal to 21 mm Hg at baseline.
7. abnormalities of the anterior segment or media opacities that prevent the assessment of the posterior segment of te eye
8. The treatment with corticosteroids (systemic, periocular or intravitreal) from at least 3 months.
9. The use of any topical medication other than the study drug for the treatment of ocular pathologies.
10. Presence or history of any systemic or ocular disease or condition that may significantly limit of visual acuity or visual field, hindering the effectiveness of treatment in the study or its evaluation, or could interfere with the interpretation of The study results, or may be judged by the investigator incompatible with the visit program or with the procedures in the study.
11. Known hypersensitivity to study drug or drugs procedural.
12. Participation in another clinical study during the same period of this study or within 90 days of the screening visit / baseline.
13. History of drug use, illegal drugs or alcohol abuse or addiction.
14. Women of childbearing potential are excluded from participation in the study if they meet one of the following conditions:

    * currently pregnant or,
    * have a positive urine pregnancy test at screening / baseline or,
    * They plan to become pregnant during the treatment period of the study or,
    * They are breast-feeding or,
    * They are not available to use highly effective measures of birth control, such as: the oral hormonal contraceptives and / or mechanical barrier methods - spermicide in conjunction with a barrier such as a condom or diaphragm or during the 'entire course of the study and 30 days after treatment periods provided.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-05; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
macular thickness | 28 days of treatment
  assessed by ocular coherence tomography (OCT)

SECONDARY OUTCOMES:
visual field | 28 days of treatment, 1 month, 6 months and 12 months of follow-up
  mean deviation
macular photoreceptors thickness | 28 days of treatment, 1 month,3 months, 6 months and 12 months of follow-up
  assessed by OCT
macular thickness | 1 month,3 months, 6 months and 12 months of follow-up
  assessed by OCT
electroretinogram (ERG) | 28 days of treatment, 1 month, 6 months and 12 months of follow-up
  amplitudes
visual acuity | 28 days of treatment,1 month,3 months, 6 months and 12 months of follow-up
contrast sensitivity | 28 days of treatment, 1 month,3 months, 6 months and 12 months of follow-up
quality of life | 28 days of treatment, 1 month,3 months, 6 months and 12 months of follow-up
number of cystoid macular edema relapses | through study completion, up to 12 months of follow-up
number of drop out for inefficacy of the study treatment | through study completion, up to 12 months of follow-up
adverse events | through study completion, up to 12 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Rama, MD, Principal Investigator — Ospedale San Raffaele. Milan
Locations (2):
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Ospedale Sacco, Milan